CLINICAL TRIAL: NCT01994330
Title: Severe Aortic Stenosis and Acquired Von Willebrand´s Disease: The Impact of Desmopressin in Valve-Replacement Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, MPoblete, Anesthesiologist, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVA
Record Dates: First submitted 2013-11-14; First posted 2013-11-25 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Acquired Von Willebrand Disease Secondary to Severe Aortic Stenosis; Heye´s Syndrome; Severe Aortic Stenosis
Keywords: acquired von Willebrand disease; severe aortic stenosis; Heye´s syndrome; desmopressin; von Willebrand multimers
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desmopressin (Experimental): 0,3 mcg per kilogram of desmopressin in 100 ml of saline, labeled as "study drug" and administered in 30 minutes a half hour before surgical incision
  Interventions: Drug: desmopressin
- placebo (Placebo Comparator): 100 of saline labeled as "study drug" administered in 30 minutes a half hour before surgical incision
  Interventions: Drug: desmopressin

INTERVENTIONS:
Drug: desmopressin — 0.3 mcg per kilogram administered in 30 minutes a half hour previous to surgical incision
  Other Names: DDAVP

SUMMARY:
Acquired Von Willebrand disease (type 2A) has been described in patients with severe aortic stenosis, the association of aortic stenosis and Digestive bleeding due to this phenomena has received the name of Heye´s syndrome.

We propose that administering Desmopressin (DDAVP) in patients scheduled to aortic valve replacement surgery will reduce blood loss and transfusion rate.

this was a pilot study

DETAILED DESCRIPTION:
Randomized Controlled trial compared with placebo in a double blind fashion. Subjects with severe aortic stenosis (transvalvular gradient >50 mmHg or valvular area of lass than 1 cm2) scheduled for aortic valve replacement were enrolled.

the day of surgery blood samples were taken in order to confirm diagnosis (factor VIII activity and Protein electrophoresis for Von Willebrand´s multimers) and then 0,3 mcg/k of DDAVP or saline equally labeled as "study drug" were administered en 30 minutes a half hour before incision.

Blood loss, postoperative hematocrit and transfusion requirement were measured, plasma sodium was measured as a safety issue.

ELIGIBILITY:
Inclusion Criteria:

* severe aortic stenosis defined as mean transvalvular gradient greater or equal to 40 mmHg ot transvalvular area less than 1 cm2
* scheduled for aortic valve replacement surgery

Exclusion Criteria:

* combined surgery (plus coronary artery bypass graft or other valve replacement/plasty)
* Infective Endocarditis
* previously known haemostatic disorder
* previous treatment with oral anticoagulants or IIb-IIIa inhibitors (we did not exclude those on acetyl-salicylic acid)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
blood loss | once patient arrives to post anesthesia care unit (approximately 6 hours after drug administration
  Blood loss obtained from fluid balance of surgery plus drain output

SECONDARY OUTCOMES:
postoperative hematocrit | the morning after surgery (18-24 hours after drug administration)
  hematocrit and hemoglobin in time frame mentioned
need of transfusion | 48 hours post administration
  transfusion of packaged red cells units until 48 hours after administration of study drug

OTHER OUTCOMES:
incidence of hyponatremia | 18-24 hours post administration of study drug
  blood sampling for plasma sodium in specified time frame
von Willebrand study and protein electrophoresis | the day of surgery, half hour previous to administration of study drug
  blood sampling for von Willebrand study:
  * collagen binding activity
  * ristocetin factor test
  * coagulation factor VIII activity
  * von Willebrand factor antigen
  * Ristocetin cofactor test/von Willebrand factor antigen ratio and protein electrophoresis of von Willebrand multimers

CONTACTS AND LOCATIONS:
Overall Officials: esperanza carrasco, anesthesiologist, Principal Investigator — Pontificia Universidad Catolica de Chile; rodrigo lopez, anesthesiologist, Study Director — Pontificia Universidad Catolica de Chile; guillermo lema, profesor titular, Study Chair — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital Clínico Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile